CLINICAL TRIAL: NCT04874896
Title: Influence of the Intestinal Microbiota on the Clinical Course of Renal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Microbiota TX (010-20)
Record Dates: First submitted 2021-04-06; First posted 2021-05-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-05

CONDITIONS: Renal Transplant

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, intervention pilot study with a sample size of 50 patients (25 patients in intervention group who will receive gut microbiota autotransplantation and 25 group in control group without intervention) for a follow-up time of 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients of this branch will not have autotransplantation of gut microbiota in capsules and will follow their usual post-transplant treatment
  Interventions: Dietary Supplement: Control
- Microbiota autotransplantation (Active Comparator): Patients in this branch will receive autotransplantation of intestinal microbiota in capsules for 6 months post-transplantation
  Interventions: Dietary Supplement: Microbiota autotransplantation

INTERVENTIONS:
Dietary Supplement: Microbiota autotransplantation — Patients received microbiota autotransplantation in capsules (1g per day) for 6 months
  Arms: Microbiota autotransplantation
Dietary Supplement: Control — Patients will not received microbiota autotransplantation in capsules and will received usual medical care
  Arms: Control

SUMMARY:
ACKGROUND: The development of new molecular techniques, in recent years, has increasing the knowledge of the composition and functionality of the intestinal microbiota. In the area of kidney transplantation, observational studies have described a change in the intestinal microbiota during the immediate post-transplantation period that seems to be related to the appearance of clinical outcomes such as diarrhea, repeated urinary tract infections, the need for adjustment of immunosuppressive treatment or acute rejection. However, intervention studies on this subject are necessary to determine how far the microbiota can influence in the development of these events.

OBJECTIVE: To clarify the influence of maintaining the composition and functionality of the intestinal microbiota on post-transplant clinical outcomes such as diarrhea, urinary tract infections, kidney graft rejection and the need for dose adjustment of immunosuppressive therapy.

MATERIALS AND METHODS: single-center, randomized, interventional pilot study with 50 deceased kidney donor transplant patients at low immunological risk. Each patient will be randomized at the time of inclusion in the study to one of the 2 branches of the study: 1) Intervention group: 25 patients who will receive a autologous fecal matter transfer during the first 6 months post-transplantation, 2) Control group: 25 renal transplant patients with the same characteristics who will not receive any type of intervention in addition to the immunosuppressive treatment indicated according to hospital protocol.

DETAILED DESCRIPTION:
ACKGROUND: The development of new molecular techniques, in recent years, has increasing the knowledge of the composition and functionality of the intestinal microbiota. In the area of kidney transplantation, observational studies have described a change in the intestinal microbiota during the immediate post-transplantation period that seems to be related to the appearance of clinical outcomes such as diarrhea, repeated urinary tract infections, the need for adjustment of immunosuppressive treatment or acute rejection. However, intervention studies on this subject are necessary to determine how far the microbiota can influence in the development of these events.

OBJECTIVE: To clarify the influence of maintaining the composition and functionality of the intestinal microbiota on post-transplant clinical outcomes such as diarrhea, urinary tract infections, kidney graft rejection and the need for dose adjustment of immunosuppressive therapy.

MATERIALS AND METHODS: single-center, randomized, interventional pilot study with 50 deceased kidney donor transplant patients at low immunological risk. Each patient will be randomized at the time of inclusion in the study to one of the 2 branches of the study: 1) Intervention group: 25 patients who will receive a autologous fecal matter transfer during the first 6 months post-transplantation, 2) Control group: 25 renal transplant patients with the same characteristics who will not receive any type of intervention in addition to the immunosuppressive treatment indicated according to hospital protocol.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of deceased donor kidney transplantation over 18 years of age, able to understand the informed consent form and who have agreed to participate in the study. Only patients with low immunological risk, whose induction for kidney transplantation was performed with basiliximab will be included, regardless of the maintenance immunosuppression combination

Exclusion Criteria:

* Recipients of deceased donor kidney transplant with high immunological risk (within the PATHI kidney transplant program).
* Kidney transplant recipients receiving pretransplant induction with thymoglobulin or polyclonal lymphocyte antiglobulin agents.
* Living donor kidney transplant recipients.
* Patients with a history of intestinal pathology such as: ulcerative colitis, Crohn's disease or malabsorptive syndrome or irritable colon prior to their inclusion in the kidney transplant waiting list.
* Patients with dysphagia, history of aspiration pneumonia or neutropenia prior to transplantation.
* Patients who, even if they meet the inclusion criteria, upon analysis of pretransplant stool, are found to be carriers of enterotoxigenic or potentially pathogenic strains such as Clostridioides difficile, or multiresistant bacteria (BLEE and/or carbapenemase-producing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the occurrence of diarrhea | 6 months after transplantation
  Evaluate the occurrence of diarrhea regardless of its cause, between the intervention and control groups. Diarrhea will be defined as three or more bowel movements per day (or more frequently than normal for the individual), and presence of loose or liquid stools, following WHO definition

SECONDARY OUTCOMES:
Occurrence of post-transplant urinary tract infections | 6 months after transplantation
  Evaluate the occurrence of post-transplant urinary tract infections (UTI), defined as positive urine culture with associated voiding symptoms or fever, as well as positive urine cultures until removal of the double J catheter, given that they will receive antibiotic treatment as if it were a UTI. Positive urine cultures or asymptomatic bacteriuria after removal of the double J catheter (usually at one-month post-transplantation) will not be included in the definition.
Evaluate the dose/level ratio of immunosuppressive drugs | 6 months after transplantation
  Evaluate the dose/level ratio of immunosuppressive drugs (tacrolimus or everolimus) administered in the intervention groups with respect to the control group
Evaluate the proportion of acute rejection episodes | 6 months after transplantation
  Evaluate the proportion of acute rejection episodes between the two groups in the follow-up period
Determined Treg lymphocyte populations | 6 months after transplantation compared to pre transplant situation
  Evaluate whether there are differences between the Treg lymphocyte populations in peripheral blood by flow cytometry between the two groups
Systemic inflammation | 6 months after transplantation
  Measurement of inflammatory markers in serum by automated systems, such as C-reactive protein
Production of bacterial metabolites | 6 months after transplantation compared to pre transplant situation
  Determination of the short-chain fatty acids (SCFA) concentration as bacterial metabolites in feces and urine by LC-MS/MS as indicators of the functionality of the microbiota
Analysis of the bacteria composing the microbiota | 6 months after transplantation compared to pre transplant situation
  Analysis of the bacteria composing the microbiota by massive sequencing of the 16S rDNA gene

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain